CLINICAL TRIAL: NCT00139789
Title: A Multicenter, Open-label Randomized Crossover Trial to Assess Subject Preference for Kemstro™ Compared to Conventional Baclofen Tablets in Subjects With Stable Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP843
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2009-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Baclofen

INTERVENTIONS:
Drug: Kemstro

SUMMARY:
This was a multicenter, open-label, randomized, crossover trial in subjects with MS who were already taking a stable dose of baclofen (up to 80 mg/day) for spasticity. The trial was designed to assess subject preference for Kemstro or conventional baclofen. At Visit 1, subjects were screened, and if qualified, were randomly assigned to one of two following treatment sequences: Kemstro/conventional baclofen or conventional baclofen/Kemstro.

ELIGIBILITY:
Inclusion Criteria:

* stable dose of baclofen

Exclusion Criteria:

* not stable dosing

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States